CLINICAL TRIAL: NCT01306214
Title: A Phase III, Randomized, Double-blind, Placebo-controlled, Parallel Group Safety and Efficacy Study of BI 10773 (10 mg and 25 mg Administered Orally Once Daily) During 52 Weeks in Patients With Type 2 Diabetes Mellitus and Insufficient Glycemic Control on MDI Insulin Regimen Alone or With Metformin
Brief Title: Safety and Efficacy of BI 10773 as add-on to Insulin Regimen in Patients With Type 2 Diabetes Mellitus
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Collaborators: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1245.49; 2010-019968-37 (EudraCT Number: EudraCT)
Record Dates: First submitted 2011-02-28; First posted 2011-03-01 (Estimated); Results first posted 2014-06-17 (Estimated); Last update posted 2014-06-17 (Estimated); Status verified 2014-05

CONDITIONS: Diabetes Mellitus, Type 2; Obesity
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Obesity | interventions — empagliflozin

ARMS (3):
- BI 10773 low dose (Experimental): BI 10773 low dose once daily
  Interventions: Drug: Placebo; Drug: BI 10773
- BI 10773 high dose (Experimental): BI 10733 high dose once daily
  Interventions: Drug: Placebo; Drug: BI 10773
- Placebo (Placebo Comparator): Placebo tablets matching BI 10773
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Placebo — Placebo matching BI 10773 low dose
  Arms: Placebo
Drug: Placebo — Placebo matching BI 10773 low dose
  Arms: BI 10773 high dose
Drug: Placebo — Placebo matching BI 10773 high dose
  Arms: Placebo
Drug: Placebo — Placebo matching BI 10773 high dose
  Arms: BI 10773 low dose
Drug: BI 10773 — BI 10773 low dose once daily
  Arms: BI 10773 low dose
Drug: BI 10773 — BI 10773 high dose once daily
  Arms: BI 10773 high dose

SUMMARY:
This trial will evaluate use of BI 10773 as add-on to insulin regimen alone or with metformin in patients with typr 2 diabetes. Both lowering glucose and HbA1c and reducing the use of insulin in this population would provide significant new information for the BI 10773 use and would offer a potential new therapeutic option in this population.

ELIGIBILITY:
Inclusion criteria:

1. Diagnosis of T2DM prior to informed consent
2. Male and female patients on diet and exercise regimen who are pre-treated with multiple daily injections (MDI) of insulin alone or in combination with immediate or extended release metformin
3. Stable metformin therapy: daily dose >=1500 mg/day or maximum tolerated dose
4. HbA1c >=7.5% and <=10% at screening

Exclusion criteria:

1. Uncontrolled hyperglycemia with a glucose level >240 mg/dl (>13.3 mmol/L) after an overnight fast during placebo run-in
2. Any contraindications to metformin according to the local label
3. Acute coronary syndrome, stroke or TIA within 3 months prior to informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 566 (Actual)
Dates: Start 2011-02; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (103):
- United States (26):
  - 1245.49.10005 Boehringer Ingelheim Investigational Site, Birmingham, Alabama
  - 1245.49.10011 Boehringer Ingelheim Investigational Site, Chandler, Arizona
  - 1245.49.10004 Boehringer Ingelheim Investigational Site, Tucson, Arizona
  - 1245.49.10002 Boehringer Ingelheim Investigational Site, Corona, California
  - 1245.49.10013 Boehringer Ingelheim Investigational Site, El Cajon, California
  - 1245.49.10030 Boehringer Ingelheim Investigational Site, Lomita, California
  - 1245.49.10014 Boehringer Ingelheim Investigational Site, Spring Valley, California
  - 1245.49.10019 Boehringer Ingelheim Investigational Site, Westlake Village, California
  - 1245.49.10024 Boehringer Ingelheim Investigational Site, Denver, Colorado
  - 1245.49.10018 Boehringer Ingelheim Investigational Site, Hialeah, Florida
  - 1245.49.10016 Boehringer Ingelheim Investigational Site, Miami, Florida
  - 1245.49.10021 Boehringer Ingelheim Investigational Site, Blue Ridge, Georgia
  - 1245.49.10009 Boehringer Ingelheim Investigational Site, Chicago, Illinois
  - 1245.49.10015 Boehringer Ingelheim Investigational Site, Evansville, Indiana
  - 1245.49.10023 Boehringer Ingelheim Investigational Site, Greenville, North Carolina
  - 1245.49.10007 Boehringer Ingelheim Investigational Site, Fargo, North Dakota
  - 1245.49.10006 Boehringer Ingelheim Investigational Site, Columbus, Ohio
  - 1245.49.10025 Boehringer Ingelheim Investigational Site, Greer, South Carolina
  - 1245.49.10022 Boehringer Ingelheim Investigational Site, Memphis, Tennessee
  - 1245.49.10003 Boehringer Ingelheim Investigational Site, Austin, Texas
  - 1245.49.10001 Boehringer Ingelheim Investigational Site, Dallas, Texas
  - 1245.49.10031 Boehringer Ingelheim Investigational Site, Houston, Texas
  - 1245.49.10033 Boehringer Ingelheim Investigational Site, Bountiful, Utah
  - 1245.49.10032 Boehringer Ingelheim Investigational Site, Salt Lake City, Utah
  - 1245.49.10026 Boehringer Ingelheim Investigational Site, Norfolk, Virginia
  - 1245.49.10020 Boehringer Ingelheim Investigational Site, Renton, Washington
- Belgium (6):
  - 1245.49.32010 Boehringer Ingelheim Investigational Site, Bonheiden
  - 1245.49.32002 Boehringer Ingelheim Investigational Site, Edegem
  - 1245.49.32007 Boehringer Ingelheim Investigational Site, Huy
  - 1245.49.32014 Boehringer Ingelheim Investigational Site, Jette
  - 1245.49.32013 Boehringer Ingelheim Investigational Site, La Louvière
  - 1245.49.32012 Boehringer Ingelheim Investigational Site, Leuven
- Bulgaria (3):
  - 1245.49.59003 Boehringer Ingelheim Investigational Site, Pleven
  - 1245.49.59004 Boehringer Ingelheim Investigational Site, Sofia
  - 1245.49.59001 Boehringer Ingelheim Investigational Site, Stara Zagora
- Colombia (5):
  - 1245.49.57003 Boehringer Ingelheim Investigational Site, Barranquilla
  - 1245.49.57004 Boehringer Ingelheim Investigational Site, Bogotá
  - 1245.49.57005 Boehringer Ingelheim Investigational Site, Bogotá
  - 1245.49.57006 Boehringer Ingelheim Investigational Site, Bogotá
  - 1245.49.57002 Boehringer Ingelheim Investigational Site, Medellín
- Czechia (6):
  - 1245.49.42003 Boehringer Ingelheim Investigational Site, Brno
  - 1245.49.42010 Boehringer Ingelheim Investigational Site, Brno
  - 1245.49.42013 Boehringer Ingelheim Investigational Site, Břeclav
  - 1245.49.42011 Boehringer Ingelheim Investigational Site, Chrudim
  - 1245.49.42009 Boehringer Ingelheim Investigational Site, Hodonín
  - 1245.49.42012 Boehringer Ingelheim Investigational Site, Svitavy56802
- Finland (3):
  - 1245.49.72001 Boehringer Ingelheim Investigational Site, Kuopio
  - 1245.49.72002 Boehringer Ingelheim Investigational Site, Oulu
  - 1245.49.72003 Boehringer Ingelheim Investigational Site, Turku
- France (9):
  - 1245.49.33001 Boehringer Ingelheim Investigational Site, Grenoble
  - 1245.49.33011 Boehringer Ingelheim Investigational Site, Le Creusot
  - 1245.49.33012 Boehringer Ingelheim Investigational Site, Marseille
  - 1245.49.33003 Boehringer Ingelheim Investigational Site, Nantes
  - 1245.49.33010 Boehringer Ingelheim Investigational Site, Narbonne
  - 1245.49.33004 Boehringer Ingelheim Investigational Site, Pierre-Bénite
  - 1245.49.33007 Boehringer Ingelheim Investigational Site, Point-à-Pitre Cedex
  - 1245.49.33008 Boehringer Ingelheim Investigational Site, Saint-Priest-en-Jarez
  - 1245.49.33009 Boehringer Ingelheim Investigational Site, Vénissieux
- Germany (6):
  - 1245.49.49104 Boehringer Ingelheim Investigational Site, Bosenheim
  - 1245.49.49013 Boehringer Ingelheim Investigational Site, Dresden
  - 1245.49.49101 Boehringer Ingelheim Investigational Site, Mainz
  - 1245.49.49002 Boehringer Ingelheim Investigational Site, Neuwied
  - 1245.49.49005 Boehringer Ingelheim Investigational Site, Saarbrücken
  - 1245.49.49102 Boehringer Ingelheim Investigational Site, Wangen
- Guatemala (5):
  - 1245.49.50201 Boehringer Ingelheim Investigational Site, Guatemala City
  - 1245.49.50202 Boehringer Ingelheim Investigational Site, Guatemala City
  - 1245.49.50203 Boehringer Ingelheim Investigational Site, Guatemala City
  - 1245.49.50204 Boehringer Ingelheim Investigational Site, Guatemala City
  - 1245.49.50205 Boehringer Ingelheim Investigational Site, Quetzaltenango
- Mexico (11):
  - 1245.49.52011 Boehringer Ingelheim Investigational Site, Aguascalientes
  - 1245.49.52012 Boehringer Ingelheim Investigational Site, Cuautla
  - 1245.49.52003 Boehringer Ingelheim Investigational Site, Durango
  - 1245.49.52005 Boehringer Ingelheim Investigational Site, Durango
  - 1245.49.52004 Boehringer Ingelheim Investigational Site, Guadalajara
  - 1245.49.52006 Boehringer Ingelheim Investigational Site, Guadalajara
  - 1245.49.52008 Boehringer Ingelheim Investigational Site, Guadalajara
  - 1245.49.52001 Boehringer Ingelheim Investigational Site, México, D.F.
  - 1245.49.52002 Boehringer Ingelheim Investigational Site, Monterrey
  - 1245.49.52009 Boehringer Ingelheim Investigational Site, Monterrey
  - 1245.49.52010 Boehringer Ingelheim Investigational Site, Monterrey
- Peru (6):
  - 1245.49.51002 Boehringer Ingelheim Investigational Site, Arequipa
  - 1245.49.51006 Boehringer Ingelheim Investigational Site, Arequipa
  - 1245.49.51010 Boehringer Ingelheim Investigational Site, Jesus Maria
  - 1245.49.51001 Boehringer Ingelheim Investigational Site, Lima
  - 1245.49.51008 Boehringer Ingelheim Investigational Site, Lima
  - 1245.49.51009 Boehringer Ingelheim Investigational Site, Lima
- Russia (4):
  - 1245.49.70008 Boehringer Ingelheim Investigational Site, Moscow
  - 1245.49.70009 Boehringer Ingelheim Investigational Site, Moscow
  - 1245.49.70006 Boehringer Ingelheim Investigational Site, Saint Petersburg
  - 1245.49.70010 Boehringer Ingelheim Investigational Site, Saint Petersburg
- Spain (8):
  - 1245.49.34039 Boehringer Ingelheim Investigational Site, Ávila
  - 1245.49.34038 Boehringer Ingelheim Investigational Site, Madrid
  - 1245.49.34044 Boehringer Ingelheim Investigational Site, Madrid
  - 1245.49.34043 Boehringer Ingelheim Investigational Site, MBoadilla Del Monte (Madrid)
  - 1245.49.34047 Boehringer Ingelheim Investigational Site, Palma de Mallorca
  - 1245.49.34045 Boehringer Ingelheim Investigational Site, Pozuelo de Alarcón
  - 1245.49.34016 Boehringer Ingelheim Investigational Site, Santiago de Compostela (La Coruña)
  - 1245.49.34041 Boehringer Ingelheim Investigational Site, Valencia
- Ukraine (5):
  - 1245.49.75016 Boehringer Ingelheim Investigational Site, Kharkiv
  - 1245.49.75007 Boehringer Ingelheim Investigational Site, Kiev
  - 1245.49.75014 Boehringer Ingelheim Investigational Site, Kiev
  - 1245.49.75015 Boehringer Ingelheim Investigational Site, Kiev
  - 1245.49.75013 Boehringer Ingelheim Investigational Site, Kyiv

REFERENCES:
- [Derived] Tuttle KR, Levin A, Nangaku M, Kadowaki T, Agarwal R, Hauske SJ, Elsasser A, Ritter I, Steubl D, Wanner C, Wheeler DC. Safety of Empagliflozin in Patients With Type 2 Diabetes and Chronic Kidney Disease: Pooled Analysis of Placebo-Controlled Clinical Trials. Diabetes Care. 2022 Jun 2;45(6):1445-1452. doi: 10.2337/dc21-2034. PMID 35472672
- [Derived] Rosenstock J, Jelaska A, Frappin G, Salsali A, Kim G, Woerle HJ, Broedl UC; EMPA-REG MDI Trial Investigators. Improved glucose control with weight loss, lower insulin doses, and no increased hypoglycemia with empagliflozin added to titrated multiple daily injections of insulin in obese inadequately controlled type 2 diabetes. Diabetes Care. 2014 Jul;37(7):1815-23. doi: 10.2337/dc13-3055. Epub 2014 Jun 14. PMID 24929430

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: Placebo matching empagliflozin 10 mg tablet plus placebo matching empagliflozin 25 mg tablet once daily
- Empagliflozin 10 mg: Empagliflozin film-coated 10 mg tablet plus one placebo matching empagliflozin 25 mg tablet once daily
- Empagliflozin 25 mg: Empagliflozin film-coated 25 mg tablet plus one placebo matching empagliflozin 10 mg tablet once daily
Period: Overall Study
Arm/Group | Placebo | Empagliflozin 10 mg | Empagliflozin 25 mg
Started | 189 | 187 | 190
Completed | 161 | 159 | 168
Not Completed | 28 | 28 | 22
Not completed — Death | 0 | 0 | 1
Not completed — Lost to Follow-up | 3 | 5 | 4
Not completed — Withdrawal by Subject | 24 | 22 | 16
Not completed — Not treated | 1 | 1 | 1

BASELINE CHARACTERISTICS:
Population: Full Analysis Set (FAS): FAS included all randomised and treated patients who had a baseline HbA1c value.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Empagliflozin 10 mg | Empagliflozin 25 mg | Total
Number analyzed (Participants) | 188 | 186 | 189 | 563
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.3 (10.1) | 56.7 (8.7) | 58.0 (9.4) | 56.7 (9.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 113 | 89 | 105 | 307
  Male | 75 | 97 | 84 | 256

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in HbA1c After 18 Weeks of Treatment
Description: The primary endpoint was the change from baseline in HbA1c after 18 weeks of treatment.
Time Frame: Baseline and 18 weeks
Population: The analysis was conducted on the full analysis set (FAS) of patients. Values after start of antidiabetic rescue therapy (week 18 definition) were set to missing and last observation carried forward (LOCF-18) was used for imputation of missing values.
Measure: Least Squares Mean (Standard Error); unit: percentage of HbA1c
Arm/Group | Placebo | Empagliflozin 10 mg | Empagliflozin 25 mg
Number analyzed (Participants) | 188 | 186 | 189
percentage of HbA1c | -0.50 (0.05) | -0.94 (0.05) | -1.02 (0.05)
Statistical Analysis 1: Comparison: Placebo vs Empagliflozin 10 mg; For the primary endpoint, the testing of the superiority hypothesis versus placebo was: Hypothesis test: H0: No difference in change from baseline to Week 18 in HbA1c (%) between Empagliflozin 10 mg and placebo Ha: A difference in change from baseline to Week 18 in HbA1c (%) between Empagliflozin 10 mg and placebo; Test type: Superiority or Other; p < 0.0001, ANCOVA — Hierarchical testing to adjust for multiple comparisons within each dose level, alpha split equally between the doses (2.5%). Empagliflozin versus placebo change from baseline in HbA1c at week 18 was the first step in each hierarchical sequence; ANCOVA Model includes baseline HbA1c as a covariate and baseline eGFR, geographic region, baseline background medication, treatment as fixed effects; Adjusted mean difference = -0.44, 97.5% CI 2-sided [-0.61 to -0.27], Standard Error of Mean 0.08 — Estimated value = Adjusted mean of Empagliflozin 10 mg - Adjusted mean of placebo
Statistical Analysis 2: Comparison: Placebo vs Empagliflozin 25 mg; For the primary endpoint, the testing of the superiority hypothesis versus placebo was: H0: No difference in change from baseline to Week 18 in HbA1c (%) between Empagliflozin 25 mg and placebo Ha: A difference in change from baseline to Week 18 in HbA1c (%) between Empagliflozin 25 mg and placebo; Test type: Superiority or Other; p < 0.0001, ANCOVA — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]; Adjusted mean difference = -0.52, 97.5% CI 2-sided [-0.69 to -0.35], Standard Error of Mean 0.07 — Estimated value = Adjusted mean of Empagliflozin 25 mg - Adjusted mean of placebo

2. Secondary Outcome: Change From Baseline in Insulin Dose After 52 Weeks of Treatment
Description: The secondary endpoint is change from baseline in insulin dose after 52 weeks of treatment
Time Frame: Baseline and 52 weeks
Population: Per Protocol Set-patients in FAS without important protocol violations leading to exclusion, completed minimum treatment of 357 days and did not prematurely discontinue. Values after start of antidiabetic rescue therapy (week 52 definition) were set to missing and last observation carried forward (LOCF-52) was used for imputation of missing values.
Measure: Least Squares Mean (Standard Error); unit: IU/day
Arm/Group | Placebo | Empagliflozin 10 mg | Empagliflozin 25 mg
Number analyzed (Participants) | 115 | 118 | 117
IU/day | 10.16 (2.16) | 1.33 (2.13) | -1.06 (2.14)
Statistical Analysis 1: Comparison: Placebo vs Empagliflozin 10 mg; Hypothesis test: H0: No difference in change from baseline to Week 52 in insulin dose (IU/day) between Empagliflozin 10 mg and placebo Ha: A difference in change from baseline to Week 52 in insulin dose (IU/day) between Empagliflozin 10 mg and placebo; Test type: Superiority or Other; p = 0.004, ANCOVA — Hierarchical testing adjusted for multiple comparisons within each dose level, alpha split equally between the doses (2.5%). Empagliflozin versus placebo change from baseline in insulin dose at week 52 was the second step in hierarchical sequence; Model - Covariates: baseline insulin daily dose,baseline HbA1c Fixed effects: baseline eGFR, region, baseline background medication, treatment; Adjusted mean difference = -8.83, 97.5% CI 2-sided [-15.69 to -1.97], Standard Error of Mean 3.05 — Estimated value = Adjusted mean of empagliflozin 10 mg - Adjusted mean of placebo
Statistical Analysis 2: Comparison: Placebo vs Empagliflozin 25 mg; Hypothesis test: H0: No difference in change from baseline to Week 52 in insulin dose (IU/day) between Empagliflozin 25 mg and placebo Ha : A difference in change from baseline to Week 52 in insulin dose (IU/day) between Empagliflozin 25 mg and placebo; Test type: Superiority or Other; p = 0.0003, ANCOVA — [p-value comment as in outcome 2, analysis 1]; [statistical method as in outcome 2, analysis 1]; Adjusted mean difference = -11.22, 97.5% CI 2-sided [-18.09 to -4.36], Standard Error of Mean 3.05 — Estimated value = Adjusted mean of Empagliflozin 25 mg - Adjusted mean of placebo

3. Secondary Outcome: Change From Baseline in Body Weight After 52 Weeks of Treatment
Description: The secondary endpoint was the change from baseline in body weight after 52 weeks of treatment
Time Frame: Baseline and 52 weeks
Population: Per Protocol Set (PPS) - completers at week 52 - using LOCF at week 52 (LOCF-52)
Measure: Least Squares Mean (Standard Error); unit: kg
Arm/Group | Placebo | Empagliflozin 10 mg | Empagliflozin 25 mg
Number analyzed (Participants) | 115 | 119 | 118
kg | 0.44 (0.36) | -1.95 (0.36) | -2.04 (0.36)
Statistical Analysis 1: Comparison: Placebo vs Empagliflozin 10 mg; Hypothesis test: H0: No difference in change from baseline to Week 52 in body weight (kg) between Empagliflozin 10 mg and placebo Ha : A difference in change from baseline to Week 52 in body weight (kg) between Empagliflozin 10 mg and placebo; Test type: Superiority or Other; p < 0.0001, ANCOVA — Hierarchical testing adjusted for multiple comparisons within each dose level, alpha split equally between the doses (2.5%). Empagliflozin versus placebo change from baseline in body weight at week 52 was the third step in hierarchical sequence; Model includes baseline weight, baseline HbA1c as covariates and baseline eGFR, region, baseline background medication, treatment as fixed effects; Adjusted mean difference = -2.39, 97.5% CI 2-sided [-3.54 to -1.24], Standard Error of Mean 0.51 — Estimated value = Adjusted mean of empagliflozin 10 mg - Adjusted mean of placebo
Statistical Analysis 2: Comparison: Placebo vs Empagliflozin 25 mg; hypothesis test: H0: No difference in change from baseline to Week 52 in body weight (kg) between Empagliflozin 25 mg and placebo Ha: A difference in change from baseline to Week 52 in body weight (kg) between Empagliflozin 25 mg and placebo; Test type: Superiority or Other; p < 0.0001, ANCOVA — [p-value comment as in outcome 3, analysis 1]; [statistical method as in outcome 3, analysis 1]; Adjusted mean difference = -2.48, 97.5% CI 2-sided [-3.63 to -1.33], Standard Error of Mean 0.51 — Estimated value = Adjusted mean of empagliflozin 25 mg - Adjusted mean of placebo

4. Secondary Outcome: Change From Baseline in HbA1c After 52 Weeks of Treatment
Description: The secondary endpoint was the change from baseline in HbA1c after 52 weeks of treatment
Time Frame: Baseline and 52 weeks
Population: Per Protocol Set (PPS) - completers at week 52 - using LOCF at week 52 (LOCF-52)
Measure: Least Squares Mean (Standard Error); unit: percentage of HbA1c
Arm/Group | Placebo | Empagliflozin 10 mg | Empagliflozin 25 mg
Number analyzed (Participants) | 115 | 119 | 118
percentage of HbA1c | -0.81 (0.08) | -1.18 (0.08) | -1.27 (0.08)
Statistical Analysis 1: Comparison: Placebo vs Empagliflozin 10 mg; H0: Difference in change from baseline to Week 52 in HbA1c (%) between empagliflozin 10 mg and placebo >0.3 Ha: Difference in change from baseline to Week 52 in HbA1c (%) between empagliflozin 10 mg and placebo ≤0.3; Test type: Non-Inferiority or Equivalence — The non- inferiority margin was 0.3%, one-sided; p < 0.0001, ANCOVA — Hierarchical testing adjusted for multiple comparisons within each dose, alpha split between the doses (2.5%). Empagliflozin versus placebo change from baseline in HbA1c at week 52 was the 4th step (non-inferiority) and 5th step (superiority); Model includes baseline HbA1c as covariate and baseline eGFR, geographical region, baseline background medication, treatment as fixed effects; Adjusted mean difference = -0.38, 97.5% CI 2-sided [-0.62 to -0.13], Standard Error of Mean 0.11 — Estimated value = Adjusted mean of empagliflozin 10 mg - Adjusted mean of placebo
Statistical Analysis 2: Comparison: Placebo vs Empagliflozin 10 mg; Hypothesis test: H0: No difference in change from baseline to Week 52 in HbA1c (%) between Empagliflozin 10 mg and placebo Ha : A difference in change from baseline to Week 52 in HbA1c (%) between Empagliflozin 10 mg and placebo; Test type: Superiority or Other; p = 0.0005, ANCOVA — [p-value comment as in outcome 4, analysis 1]; [statistical method as in outcome 4, analysis 1]; Adjusted mean difference = -0.38, 97.5% CI 2-sided [-0.62 to -0.13], Standard Error of Mean 0.11 — Estimated value = Adjusted mean of empagliflozin 10 mg - Adjusted mean of placebo
Statistical Analysis 3: Comparison: Placebo vs Empagliflozin 25 mg; H013: Difference in change from baseline to Week 52 in HbA1c (%) between empagliflozin 25 mg and placebo >0.3 Ha13: Difference in change from baseline to Week 52 in HbA1c (%) between empagliflozin 25 mg and placebo ≤0.3; Test type: Non-Inferiority or Equivalence — The non- inferiority margin was 0.3%, one-sided; p < 0.0001, ANCOVA — [p-value comment as in outcome 4, analysis 1]; [statistical method as in outcome 4, analysis 1]; Adjusted mean difference = -0.46, 97.5% CI 2-sided [-0.70 to -0.22], Standard Error of Mean 0.11 — Estimated value = Adjusted mean of empagliflozin 25 mg - Adjusted mean of placebo
Statistical Analysis 4: Comparison: Placebo vs Empagliflozin 25 mg; Hypothesis test: H0: No difference in change from baseline to Week 52 in HbA1c (%) between Empagliflozin 25 mg and placebo Ha : A difference in change from baseline to Week 52 in HbA1c (%) between Empagliflozin 25 mg and placebo; Test type: Superiority or Other; p < 0.0001, ANCOVA — [p-value comment as in outcome 4, analysis 1]; [statistical method as in outcome 4, analysis 1]; Adjusted mean difference = -0.46, 97.5% CI 2-sided [-0.70 to -0.22], Standard Error of Mean 0.11 — Estimated value = Adjusted mean of empagliflozin 25 mg - Adjusted mean of placebo

ADVERSE EVENTS:
Time Frame: Up to 52 weeks
Description: An adverse event is defined as any untoward medical occurrence in a clinical investigation subject administered a pharmaceutical product and which does not necessarily have a causal relationship with this treatment. At each visit adverse events were recorded on a cumulative case report form.
Arm/Group | Placebo | Empagliflozin 10 mg | Empagliflozin 25 mg
Serious Adverse Events (participants affected / at risk) | 22/188 | 20/186 | 22/189
Other Adverse Events (participants affected / at risk) | 146/188 | 135/186 | 140/189
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=188) | Empagliflozin 10 mg (N=186) | Empagliflozin 25 mg (N=189)
Pneumonia (Infections and infestations) | 1 | 3 | 1
Anal abscess (Infections and infestations) | 0 | 1 | 0
Appendicitis (Infections and infestations) | 1 | 0 | 0
Diabetic gangrene (Infections and infestations) | 1 | 0 | 0
Gastrointestinal infection (Infections and infestations) | 0 | 1 | 0
Lobar pneumonia (Infections and infestations) | 0 | 0 | 1
Sepsis (Infections and infestations) | 0 | 1 | 0
Subcutaneous abscess (Infections and infestations) | 1 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 1
Ependymoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Glioblastoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Pancreatic carcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Anaemia (Blood and lymphatic system disorders) | 1 | 0 | 0
Sarcoidosis (Immune system disorders) | 0 | 1 | 0
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 1 | 0 | 0
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 1 | 1 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Depression (Psychiatric disorders) | 1 | 0 | 0
Carpal tunnel syndrome (Nervous system disorders) | 1 | 0 | 0
Cerebrovascular accident (Nervous system disorders) | 1 | 1 | 0
Cervicobrachial syndrome (Nervous system disorders) | 1 | 0 | 0
Convulsion (Nervous system disorders) | 0 | 1 | 0
Grand mal convulsion (Nervous system disorders) | 0 | 1 | 0
Migraine (Nervous system disorders) | 1 | 0 | 0
Radiculitis (Nervous system disorders) | 1 | 0 | 0
Syncope (Nervous system disorders) | 0 | 1 | 1
Amaurosis (Eye disorders) | 0 | 0 | 1
Angle closure glaucoma (Eye disorders) | 0 | 1 | 0
Pterygium (Eye disorders) | 0 | 1 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 2 | 1
Vertigo positional (Ear and labyrinth disorders) | 0 | 1 | 0
Coronary artery disease (Cardiac disorders) | 2 | 0 | 1
Acute myocardial infarction (Cardiac disorders) | 0 | 0 | 1
Angina pectoris (Cardiac disorders) | 0 | 0 | 1
Bundle branch block right (Cardiac disorders) | 1 | 0 | 0
Cardiac failure (Cardiac disorders) | 0 | 0 | 1
Cardiac failure congestive (Cardiac disorders) | 1 | 0 | 1
Cor pulmonale (Cardiac disorders) | 0 | 0 | 1
Supraventricular tachycardia (Cardiac disorders) | 1 | 0 | 0
Tachycardia (Cardiac disorders) | 0 | 1 | 0
Hypertensive emergency (Vascular disorders) | 1 | 0 | 0
Orthostatic hypotension (Vascular disorders) | 0 | 0 | 1
Peripheral arterial occlusive disease (Vascular disorders) | 0 | 0 | 1
Peripheral artery stenosis (Vascular disorders) | 0 | 0 | 1
Thrombophlebitis migrans (Vascular disorders) | 0 | 1 | 0
Venous thrombosis (Vascular disorders) | 1 | 0 | 0
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 2 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 1
Gastric ulcer (Gastrointestinal disorders) | 1 | 0 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0
Pancreatitis acute (Gastrointestinal disorders) | 0 | 0 | 1
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 1
Umbilical hernia (Gastrointestinal disorders) | 0 | 0 | 1
Diabetic foot (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Skin ulcer (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Intervertebral disc disorder (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Neuropathic arthropathy (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Acute prerenal failure (Renal and urinary disorders) | 0 | 0 | 1
Renal colic (Renal and urinary disorders) | 0 | 1 | 0
Renal failure acute (Renal and urinary disorders) | 0 | 0 | 1
Renal impairment (Renal and urinary disorders) | 0 | 1 | 0
Ectopic pregnancy (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 1
Concussion (Injury, poisoning and procedural complications) | 0 | 0 | 1
Humerus fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Wound (Injury, poisoning and procedural complications) | 0 | 1 | 0
Vitrectomy (Surgical and medical procedures) | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=188) | Empagliflozin 10 mg (N=186) | Empagliflozin 25 mg (N=189)
Nasopharyngitis (Infections and infestations) | 40 | 34 | 27
Urinary tract infection (Infections and infestations) | 23 | 24 | 24
Influenza (Infections and infestations) | 12 | 7 | 14
Bronchitis (Infections and infestations) | 12 | 10 | 8
Gastroenteritis (Infections and infestations) | 10 | 8 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 111 | 97 | 110
Hyperglycaemia (Metabolism and nutrition disorders) | 14 | 6 | 7
Dizziness (Nervous system disorders) | 2 | 5 | 13
Headache (Nervous system disorders) | 9 | 8 | 11
Hypertension (Vascular disorders) | 10 | 9 | 7
Diarrhoea (Gastrointestinal disorders) | 17 | 12 | 17
Arthralgia (Musculoskeletal and connective tissue disorders) | 10 | 18 | 11
Back pain (Musculoskeletal and connective tissue disorders) | 14 | 12 | 15

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Any publication of the result of this trial must be consistent with the Boehringer Ingelheim publication policy. The rights of the investigator and of the sponsor with regard to publication of the results of this trial are described in the investigator contract.